CLINICAL TRIAL: NCT03054220
Title: Risk of Phenoconversion in Genetic Extensive Metabolizers Healthy Volunteers Carriers of One Fully-Functional and One Non-Functional Allele Versus Carriers of Two Fully-Functional Alleles
Brief Title: Impact of Genetic Polymorphism on Drug-Drug Interactions Involving CYP2D6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Desmeules (Other)
Responsible Party: Sponsor-Investigator, Jules Desmeules, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-00262
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Dextromethorphan; Tramadol; Duloxetine Hydrochloride; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYP2D6 gene score 1 (Experimental): carriers of 1 fully functional and 1non functional CYP2D6 alleles
  Interventions: Drug: Dextromethorphan 5 MG; Drug: Tramadol 10 mg; Drug: Duloxetine 60mg; Drug: Paroxetine 20 mg
- CYP2D6 gene score 2 (Experimental): carriers of 2 fully functional CYP2D6 alleles
  Interventions: Drug: Dextromethorphan 5 MG; Drug: Tramadol 10 mg; Drug: Duloxetine 60mg; Drug: Paroxetine 20 mg

INTERVENTIONS:
Drug: Dextromethorphan 5 MG
Drug: Tramadol 10 mg
Drug: Duloxetine 60mg
Drug: Paroxetine 20 mg

SUMMARY:
CYP2D6 is characterized by a huge variability in the general population, mainly because of genetic polymorphism and drug-drug interactions (DDIs). CYP2D6 genotype is known to have an impact on the extent of DDIs. Indeed several studies have pointed out differential DDIs extent according to CYP2D6 genotype. The terms phenoconversion and phenotype switch are both used to describe the phenomenon by which a given subject changes his phenotype to another due external influence such as DDIs. When given a sufficiently strong CYP2D6 inhibitor, the phenotype of an individual with no mutant allele (extensive metabolizer, EM) of CYP2D6 can be modified to a poor metabolizer (PM) phenotype. This vulnerability is also thought to be dependent on CYP2D6 genotype. Various combinations of alleles predict an EM genotype, which represents about 60 to 70% of the general population. The aim of the study is to determine whether the presence of genetic mutation in CYP2D6 has an impact on DDIs involving the CYP2D6 enzyme. Our interest focuses on CYP2D6 EM carriers of two fully functional alleles and carriers of one non-functional and one functional allele. In order to elucidate this question, CYP2D6 activity will be measured on healthy volunteers by administration of single low doses of dextromethorphan and tramadol in presence or not of duloxetine and paroxetine, two known CYP2D6 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-60 years
* Body Mass Index 18-27
* Understanding of French language and able to give a written inform consent
* CYP2D6 genotype : combination of two fully-functional (normal activity) alleles or of one fully-functional and one non-functional allele (null activity), according to table 1, without gene multiplication

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Any pathologies, use of drugs or food that may affect CYP2D6 activity
* Regular smokers of >5 cigarettes/day
* Renal or hepatic impairment
* Medical history of chronic alcoholism or abuse of psychoactive drugs, including opiate addiction
* Liver transplantation
* Sensitivity to any of the drugs used
* Alteration of hepatic tests more than 2x normal
* Glomerular filtration rate < 60 ml/min/1.73m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Difference in the proportion of volunteers with urinary metabolic ratio Dextromethorphan/Dextrorphan >0.3 | 10 hours

SECONDARY OUTCOMES:
AUC of plasmatic concentrations probe drugs (dextromethorphan and tramadol) and their metabolites and tramadol) and their metabolites in plasma | 24 hours
Cmax of probe drugs (dextromethorphan and tramadol) and their metabolites and tramadol) and their metabolites in plasma and tramadol) and their metabolites in plasma | 24 hours
Tmax of plasmatic concentrations probe drugs (dextromethorphan and tramadol) and their metabolites and tramadol) and their metabolites in plasma and tramadol) and their metabolites in plasma | 24 hours
Half-life of probe drugs (dextromethorphan and tramadol) and their metabolites and tramadol) and their metabolites in plasma and tramadol) and their metabolites in plasma | 24 hours
Clearance of probe drugs (dextromethorphan and tramadol) and their metabolites and tramadol) and their metabolites in plasma | 24 hours
Difference in the urinary metabolic ratio tramadol/M1 | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jules A Desmeules, Pr, Principal Investigator — HUG